CLINICAL TRIAL: NCT04793126
Title: Clinical and Urodynamic Evaluation of Surgical Repair of Pelvic Organ Prolapse Associated With Lower Urinary Tract Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Gamil Ahmed Higazy, Assistant lecturer, Ain Shams University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAMSU 1743/2013
Record Dates: First submitted 2021-03-09; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: All patients were subjected to clinical evaluation and urodynamic testing before surgery. All cases underwent surgical repair of pelvic organ prolapse. Follow-up clinical examination was performed at 1, 3, and 6 months postoperatively, and urodynamic examination was repeated 6 months after repair.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Urodynamic study — comparison between the urodynamic study of the patients before pelvic prolapse surgical repair and 6 months later.

SUMMARY:
To assess the urinary symptoms and urodynamic findings concomitant with Pelvic organ prolapse before and after surgical treatment and to define the role of urodynamic study in treatment decision making.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is a prevalent problem that affects women's quality of life women with POP may present with a variety of lower urinary tract symptoms (LUTS).

For POP patients with concomitant urinary symptoms, urodynamic (UDN) testing is proposed for proper evaluation of cases and identification of the pathophysiologic events in each case individually.

In this prospective study, the investigators aim to describe the urinary symptoms and urodynamic findings concomitant with POP before and after surgical treatment of POP. We also aimed at defining the role of UDN in decision-making regarding the treatment of POP when associated with LUTS.

ELIGIBILITY:
Inclusion Criteria:

* women with anterior pelvic organ prolapse (POP) associated with Lower urinary tract symptoms

Exclusion Criteria:

* Patients with POP less than POP-Q grade II, POP not in need for surgical repair, neurological diseases that could possibly affect voiding functions, pelvic infections, congenital bladder disorders, history of urinary fistula, history of malignancy, and patients on current medical treatment for voiding dysfunction.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pelvic organ prolapse surgeries
Enrollment: 83 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Urodynamic study evaluation for the participants | 6 month after the procedure
  evaluation of the urodynamic study after the surgical repair of the pelvic organ prolapse and comparison to the preoperative results.